CLINICAL TRIAL: NCT02065908
Title: Circulating microRNAs as a Novel Biomarker of Early Cardiotoxicity in Breast Cancer Patients Treated With Anthracyclines
Brief Title: Circulating MicroRNA as Biomarker of Cardiotoxicity in Breast Cancer
Status: Completed | Type: Observational
Sponsor: West Pomeranian Cancer Center (Other)
Collaborators: Pomeranian Medical University Szczecin (Other)
Responsible Party: Principal Investigator, Bartosz Dąbek, MD, West Pomeranian Cancer Center
Other Study IDs: ZCO-2014-BD
Record Dates: First submitted 2014-02-15; First posted 2014-02-19 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-12

CONDITIONS: Breast Cancer
Keywords: breast cancer; anthracyclines; cardiotoxicity; circulating microRNA; biomarker; serum; anthracyclines based chemotherapy
MeSH Terms: conditions — Breast Neoplasms; Cardiotoxicity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 5 ml of blood will be collected, 2ml of serum will be isolated from the blood and stored below -80C till completion of the study.
Oversight: Data Monitoring Committee: No

SUMMARY:
In the proposed project the investigators will asses whether changes in expression of selected circulating microRNAs in serum could comprise a sensitive and specific biomarker of cardiotoxicity in cancer patients treated with anthracyclines based chemotherapy.

DETAILED DESCRIPTION:
Blood will be taken

1. before anthracycline based chemotherapy administration
2. at the middle of anthracycline treatment (before 3rd and/or 5th cycle of drugs infusion)
3. after anthracycline chemotherapy cessation
4. 6 months after chemotherapy cessation if an end point occurs
5. 12 months after chemotherapy cessation if an end point occurs

Echocardiography will be performed

1. before anthracycline based chemotherapy administration
2. after anthracycline based chemotherapy cessation
3. 6 months after anthracycline based chemotherapy cessation
4. 12 months after anthracycline based chemotherapy cessation if no end point was observed earlier The investigators will perform high-throughput miRNA(microRNA) expression profiling of serum samples - called training set.

Training set will consist of sera of 30 patients who has reached an end point. Training set will be sequenced using next generation sequencing.

Training set will be used to derive a miRNA signature capable of separating early cardiotoxicity patients from healthy ones. MiRNA signature will be validated using validation set.

ELIGIBILITY:
Inclusion Criteria:

* age 18-70
* stage I-III TNM (Tumor Node Metastases)

Exclusion Criteria:

* second or next cancer (except for basal cell skin cancer and CIN)
* previously treated with chemotherapy
* previously treated with radiotherapy
* acute myocardial infarction
* heart failure
* cardiomyopathy

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with newly diagnosed breast cancer that will be treated with anthracyclines will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2014-01; Primary Completion 2016-06 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Cardiotoxicity events according to CREC (Cardiac Review and evaluation Committee) criteria | up to 76 weeks after chemotherapy conclusion
  either a cardiomyopathy with decreased left ventricular ejection fraction (LVEF), a reduction of LVEF ≥5% to <55% with symptoms of heart failure (e.g. orthopnoea and paroxysmal nocturnal dyspnoea, elevated jugular venous pressure, S3 gallop, Hepatojugular reflux, tachycardia), or an asymptomatic reduction of LVEF ≥10% to <55%

CONTACTS AND LOCATIONS:
Overall Officials: Bartosz Dąbek, MD, Principal Investigator — West Pomeranian Cancer Center
Locations (3):
- Poland (3):
  - Clinical Oncology Department, West Pomeranian Cancer Center, Szczecin, West Pomeranian Voivodeship
  - Collegium Medicum of Jagiellonian University, Krakow
  - Pomeranian Medical University, Department of Cardiology, Szczecin